CLINICAL TRIAL: NCT04989426
Title: State of Health and Integration Into the Health Care System of Migrant Patients, New Arrivals, Consultants in Urban Primary Care Structures,in Seine Saint Denis and in the North of Paris.
Brief Title: Generalist Cohort of Migrant Patients Consultants in City Medicine
Acronym: CoPAMViL
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210936
Record Dates: First submitted 2021-07-19; First posted 2021-08-04 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Care System for Newly Arrived Migrants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: the state of health of newly arrived migrant patients in the year following their arrival in France — the state of health of newly arrived migrant patients in the year following their arrival in France

SUMMARY:
This innovative cross-sectional study, carried out in the city, will provide valuable prospective data that will make it possible to identify public health avenues for specific and adapted care both in the medical and social field of newcomers to our territory. Our study will characterize the impact of reforms of the conditions of access to State medical aid and universal health protection on access to care and the state of health of this population. . It will make it possible to participate in the advocacy in favor of access to healthcare for all and the city PASS, the only device allowing access to healthcare in the city for all newcomers regardless of their status.

DETAILED DESCRIPTION:
Participants will be informed orally and via an information note written by the doctor during their first medical contact in France or during a follow-up visit within the municipal health center.

The health data comes from the participant's care file and some social data is extracted from the social information system, already existing and used by the reception agents responsible for the consultations. access to rights.

Inclusion visit :

This visit will take place during the first medical visit of eligible patients.

During this visit, the investigative team:

* Checks the inclusion and non-inclusion criteria;
* Gives clear oral and written information;
* Collect the patient's non-opposition;
* Performs the medico-social consultation in accordance with the management recommendations.

Follow-up visits Follow-up will be continued 12 months after the inclusion visit. The rhythm, as well as the nature of the follow-up visits for the patients included, will be defined by the information obtained during the inclusion visit, and will be determined by the doctor in charge of the patient.

For patients included retrospectively The inclusion visit will take place during a follow-up medico-social visit planned as part of the care in one of the participating the municipal health center.

During this visit, the investigative team:

* Checks the inclusion and non-inclusion criteria;
* Gives clear oral and written information;
* Collect the patient's non-opposition;
* Performs the medico-social consultation in accordance with the management recommendations

During the inclusion visit and medical follow-up visits, within the Municipal Health Centers, a consultation on access to rights will also be carried out in order to help patients put together their social file.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥ 18 years)
* Newly arrived migrants (foreigners born outside France, first arrival in France AND presence in the territory ≤ 1 year)
* 1st medical contact in town medicine in France

Exclusion Criteria:

* Refusal of participation
* Communication impossible due to the language barrier despite translation or interpreting (telephone or face-to-face)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: specific population of major newcomer migrants
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
The number of medical and social consultations one year after inclusion. | one year after arrival in France
  describe the state of health of newly arrived migrant patients in the year following their arrival in France
Number of newcomer biological assessments prescribed by the doctor one year after inclusion | one year after arrival in France
  describe the state of health of newly arrived migrant patients in the year following their arrival in France

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CMS Aubervilliers, Aubervilliers
  - CMS Saint-Denis, Saint-Denis

IPD SHARING:
Plan to Share IPD: No
* The data will be entered in an electronic CRF: Cleanweb®, hosted in France on a health data host.
  * Allocation of an individual code to each participant eligible for the research: center number, serial number in the research, initial Last name and initial First name
  * Use of a correspondence table (kept in the center by the principal investigator until the publication of the research article)
  Non-identifying data will be entered into an electronic Cleanweb CRF and each participant will be assigned an individual code.
  The computer session and access to the e-CRF will be protected by a user code and a password.